CLINICAL TRIAL: NCT00590005
Title: Redox Determinants of Severe Asthma: A Substudy of the NHLBI Severe Asthma Research Program
Brief Title: Redox Determinants of Severe Asthma (a Substudy of the Severe Asthma Research Program)
Acronym: SARP
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Collaborators: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Anne M Fitzpatrick PhD, Assistant Professor, Emory University
Other Study IDs: IRB00024906; 2R01HL069170-07 (NIH)
Record Dates: First submitted 2007-12-27; First posted 2008-01-10 (Estimated); Results first posted 2014-01-13 (Estimated); Last update posted 2014-02-10 (Estimated); Status verified 2014-01

CONDITIONS: Asthma
Keywords: severe asthma; poorly controlled asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Children with severe asthma: This group consists of children with severe asthma as defined per ATS workshop criteria (published in 2000).
- Children with non-severe asthma: This group includes children with asthma who do not meet the ATS criteria for severe asthma as outlined in the 2000 workshop report.

SUMMARY:
Hypotheses: 1) Airway pH regulation is abnormal in severe asthma; 2) In severe asthma, there is formation of cytotoxic nitrogen oxides and loss of beneficial nitrogen oxides in the airways

DETAILED DESCRIPTION:
Specific Aim 1:Test hypothesis that airway pH regulation is abnormal in severe asthma.

1a) Determine the effects of systemic corticosteroids on breath pH in children with severe and mild to moderate asthma.

1b) Examine whether breath condensate pH and other biomarkers of oxidant stress can predict clinical outcomes in children with severe and mild to moderate asthma.

1c) Identify whether increased Th1/Th2 cytokine ratio, and abnormalities in airway glutaminase, G-SNO-reductase, VATPase, and carbonic anhydrase are associated with airway pH disturbance in children with severe asthma.

1d) Test whether rhinovirus infections, which reduce airway pH, persist longer or are more frequent in children with severe asthma than in children with mild to moderate asthma.

1e) Examine the relationship between gastroesophageal reflux and proximal airway pH in children with severe asthma and mild to moderate asthma.

ELIGIBILITY:
Inclusion Criteria:

* At least 6 years old
* Asthma diagnosis by physician
* Current treatment with an inhaled corticosteroid medication

Exclusion criteria:

* Bronchiectasis
* Cystic Fibrosis
* Chronic Obstructive Pulmonary Disease

Ages: 6 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study population consists of children with physician-diagnosed asthma in the Atlanta, Georgia area across a wide range of asthma severities (mild, moderate, severe)
Sampling Method: Non-Probability Sample
Enrollment: 225 (Actual)
Dates: Start 2003-01; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: W G Teague, MD, Principal Investigator — University of Virginia
Locations (1):
- Emory Childrens Center, Atlanta, Georgia, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Children were recruited from January 2003 to June 2011 from the Emory Children's Center asthma clinic.
Pre-assignment Details: Children with physician diagnosed asthma were enrolled and underwent comprehensive phenotypic characterization consisting of pulmonary function measures, biomarker assessment, and allergy assessment.
Groups:
- Children With Severe Asthma: This group includes children with severe asthma diagnosed according to American Thoracic Society criteria (2000 workshop definition)
- Children With Non-severe Asthma: This group includes child with physician-diagnosed asthma who did not meet criteria for severe asthma.
Period: Overall Study
Arm/Group | Children With Severe Asthma | Children With Non-severe Asthma
Started | 106 | 119
Completed | 106 | 119
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Children With Asthma: The cohort consists of children with physician-diagnosed asthma across a wide range of severity (mild, moderate, severe)
Arm/Group | Children With Asthma
Number analyzed (Participants) | 225
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 225
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.8 (3.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 102
  Male | 123
Region of Enrollment [Number; unit: participants]
  United States | 225

OUTCOME MEASURES:

1. Primary Outcome: Exhaled Nitric Oxide at Baseline and Over the Observational Period
Description: Exhaled nitric oxide concentrations as measured by collection of exhaled breath into a mylar bag
Time Frame: baseline and after 21 days
Population: 225 children were enrolled into the study and completed baseline assessments. Only 40 children were followed longitudinally. The results from only those 40 children are shown here.
Measure: Mean (Standard Deviation); unit: parts per billion
Arm/Group | Children With Severe Asthma | Children With Non-severe Asthma
Number analyzed (Participants) | 20 | 20
parts per billion
  Exhaled nitric oxide value at 21 days | 15.1 (5.4) | 9.9 (5.8)
  Exhaled nitric oxide baseline value | 13.7 (7.4) | 8.6 (6.2)

2. Secondary Outcome: Reduction in Breath pH
Description: Breath condensate pH was measured by the RTube (trademark) device. This device is a plastic tube with a one-way exhalation valve and a chilled aluminum sleeve. pH (the log of hydrogen ion concentration) was measured using an Orion pH meter and probe calibrated in 4.0, 7.0, and 10.0 pH solutions.
Time Frame: baseline and 21 days
Population: 225 children with asthma were enrolled in the study and completed baseline assessments. Only 40 children were followed longitudinally. The data from those 40 children are shown here.
Measure: Mean (Standard Deviation); unit: log of hydrogen ion concentration (pH)
Arm/Group | Children With Severe Asthma | Children With Non-severe Asthma
Number analyzed (Participants) | 20 | 20
log of hydrogen ion concentration (pH)
  Breath pH at 21 days | 7.08 (0.52) | 7.58 (0.32)
  Breath pH at baseline | 7.68 (0.69) | 7.63 (0.88)

ADVERSE EVENTS:
Time Frame: adverse event data were collected for 3 months.
Arm/Group | Children With Severe Asthma | Children With Non-severe Asthma
Serious Adverse Events (participants affected / at risk) | 0/106 | 0/119
Other Adverse Events (participants affected / at risk) | 0/106 | 0/119

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No